CLINICAL TRIAL: NCT03670316
Title: Effectiveness of a Smoking Cessation Algorithm Integrated Into HIV Primary Care
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University of Washington (Other); Harvard University (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Karen Cropsey, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 300000632; R01DA044112 (NIH)
Record Dates: First submitted 2018-09-05; First posted 2018-09-13 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: HIV; AIDS; Smoking Cessation
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Smoking Cessation

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either the Algorithm Treatment plus referral to a quitline (AT) or the quitline alone condition (eTAU).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Algorithm Treatment plus referral to quitline (AT) (Experimental): will be assigned a pharmacotherapy treatment regimen recommended to their provider.
  Interventions: Drug: Algorithm Treatment
- Quitline (eTAU) (Active Comparator): will be referred to quitlines, telephone-based tobacco cessation services.
  Interventions: Other: Quitline only

INTERVENTIONS:
Drug: Algorithm Treatment — Varenicline was selected as the first line of treatment for patients willing to take a medication twice per day and wanting cessation. Following varenicline, bupropion and then NRT are subsequent options. In terms of preference for NRT, nicotine patches would be the first option followed by lozenge, gum, inhaler, and nasal spray. The order of NRT within the algorithm is based upon patient familiarity and number of clinical trials supporting their use. Combination NRT (e.g., patch and lozenge) or adding NRT to varenicline or bupropion is offered to participants who have made an unsuccessful quit attempt with these medications in the past. If none of these medications are appropriate, then the participant is offered counseling only.
  Arms: Algorithm Treatment plus referral to quitline (AT)
Other: Quitline only — eTAU participants will complete the same algorithm questions but will not have this information sent to their provider, although their provider may elect to prescribe medication as part of standard of care. Participants will be referred to a quitline for behavioral support services for cessation.
  Arms: Quitline (eTAU)

SUMMARY:
To determine the efficacy of an algorithm designed to recommend smoking cessation-related pharmacotherapy options to the primary care providers of smokers living with HIV/AIDS.

DETAILED DESCRIPTION:
Smoking remains the leading cause of preventable death and disability in the United States. Whereas smoking has declined significantly among individuals in the general population, it is clustered in populations of vulnerable individuals such as people living with HIV/AIDS (PLWH) in whom smoking prevalence rates and resulting comorbidity rates remain high. Medical advances in the treatment of HIV have resulted in substantial increases in life expectancy among PLWH and as a consequence PLWH smokers are now, more than ever, at heightened risk for tobacco-related illnesses and death. PLWH smokers engaged in treatment lose more years of life due to smoking now than to HIV disease. Although PLWH smokers engaged in HIV care typically see a medical provider every 4-6 months, smoking cessation treatment and referral is often not part of routine HIV care. While 94% of HIV treatment providers indicated that they would be willing to provide smoking cessation services to their patients, few have received training in how to provide smoking cessation services. With seven first line pharmacotherapies available for smoking cessation, development of algorithms to assist providers in selecting the most appropriate pharmacotherapy is an important but untested strategy to increase smoking cessation in PLWH. The purpose of this proposal is to conduct a mixed efficacy/effectiveness trial comparing an algorithm treatment with prescription cost off sets and quit line referral (AT) to an enhanced Treatment as Usual (quit line referral only; eTAU) group. Six hundred PLWH smokers will be recruited at the University of Alabama at Birmingham, University of Washington, and Fenway Health HIV clinics and will be randomized to receive AT or eTAU. All AT smokers will receive active treatment for twelve weeks regardless of stated motivation or intention to quit. eTAU smokers will be referred to quit line services and HIV providers may elect to treat smoking as part of standard of care. Participants will remain in the study for 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Enrollment in the CNICS clinical cohort.
2. 18 years or older;
3. Receiving HIV care at the UAB, UW or Fenway Health clinics and not anticipating changing clinics over the next six months
4. Smoking greater than or equal to 5 cigarettes per day (cpd) for the past month
5. Living in an unrestricted environment that allows smoking.

Exclusion Criteria:

1. Cognitive impairment such that unable to provide informed consent;
2. Non-English speaking;
3. Acutely suicidal, manic, acutely intoxicated, or otherwise not stable enough to provide informed consent;
4. Currently receiving smoking cessation treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
7-day point-prevalence abstinence | 6 months
  Number of cigarettes smoked over the past 7 days

SECONDARY OUTCOMES:
Cigarettes per day | 6 months
  Number of cigarettes reported being smoked per day
24 hour quit attempts | 6 months
  Attempt to not smoke for 24 hours
Number of prescriptions written | 6 months
  The number of prescriptions written for a participant

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama, Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Background] Seger, J. C., Horn, D. B., Westman, E. C., Lindquist, R., Scinta, W., Richardson, L. A., ... & Bays, H. E. (2013). American Society of Bariatric Physicians Obesity Algorithm: Adult Adiposity Evaluation and Treatment 2013.
- [Background] Barst RJ, Gibbs JSR, Ghofrani HA, Hoeper MM, McLaughlin VV, Rubin LJ, Sitbon O, Tapson VF, Galie N. Updated evidence-based treatment algorithm in pulmonary arterial hypertension. J Am Coll Cardiol. 2009 Jun 30;54(1 Suppl):S78-S84. doi: 10.1016/j.jacc.2009.04.017. PMID 19555861
- [Background] Nathan DM, Buse JB, Davidson MB, Ferrannini E, Holman RR, Sherwin R, Zinman B; American Diabetes Association; European Association for Study of Diabetes. Medical management of hyperglycemia in type 2 diabetes: a consensus algorithm for the initiation and adjustment of therapy: a consensus statement of the American Diabetes Association and the European Association for the Study of Diabetes. Diabetes Care. 2009 Jan;32(1):193-203. doi: 10.2337/dc08-9025. Epub 2008 Oct 22. PMID 18945920
- [Background] Hughes JR. An updated algorithm for choosing among smoking cessation treatments. J Subst Abuse Treat. 2013 Aug;45(2):215-21. doi: 10.1016/j.jsat.2013.01.011. Epub 2013 Mar 19. PMID 23518288
- [Background] Hughes J. An algorithm for choosing among smoking cessation treatments. J Subst Abuse Treat. 2008 Jun;34(4):426-32. doi: 10.1016/j.jsat.2007.07.007. Epub 2007 Sep 14. PMID 17869475
- [Background] Bader P, McDonald P, Selby P. An algorithm for tailoring pharmacotherapy for smoking cessation: results from a Delphi panel of international experts. Tob Control. 2009 Feb;18(1):34-42. doi: 10.1136/tc.2008.025635. Epub 2008 Oct 9. PMID 18845621
- [Background] Kunyk D, Els C, Papadakis S, Selby P. Tobacco use disorder treatment in primary care: implementing a clinical system pathway in Alberta. Can Fam Physician. 2014 Jul;60(7):646-55. PMID 25022640
- [Background] Fiore, M. C., C. R. Jaen, et al. (2008). Treating tobacco use and dependence: 2008 Update. Clinical Practice Guideline. Rockville, MD, US Public Health Service.
- [Background] Shuter J, Bernstein SL, Moadel AB. Cigarette smoking behaviors and beliefs in persons living with HIV/AIDS. Am J Health Behav. 2012 Jan;36(1):75-85. doi: 10.5993/ajhb.36.1.8. PMID 22251785
- [Background] Schnoll RA, Rukstalis M, Wileyto EP, Shields AE. Smoking cessation treatment by primary care physicians: An update and call for training. Am J Prev Med. 2006 Sep;31(3):233-9. doi: 10.1016/j.amepre.2006.05.001. Epub 2006 Jul 24. PMID 16905034
- [Background] Aveyard P, Begh R, Parsons A, West R. Brief opportunistic smoking cessation interventions: a systematic review and meta-analysis to compare advice to quit and offer of assistance. Addiction. 2012 Jun;107(6):1066-73. doi: 10.1111/j.1360-0443.2011.03770.x. Epub 2012 Feb 28. PMID 22175545
- [Background] Carpenter MJ, Hughes JR, Gray KM, Wahlquist AE, Saladin ME, Alberg AJ. Nicotine therapy sampling to induce quit attempts among smokers unmotivated to quit: a randomized clinical trial. Arch Intern Med. 2011 Nov 28;171(21):1901-7. doi: 10.1001/archinternmed.2011.492. PMID 22123796
- [Background] Ingersoll KS, Cropsey KL, Heckman CJ. A test of motivational plus nicotine replacement interventions for HIV positive smokers. AIDS Behav. 2009 Jun;13(3):545-54. doi: 10.1007/s10461-007-9334-4. Epub 2007 Dec 8. PMID 18066659
- [Background] Lloyd-Richardson EE, Stanton CA, Papandonatos GD, Shadel WG, Stein M, Tashima K, Flanigan T, Morrow K, Neighbors C, Niaura R. Motivation and patch treatment for HIV+ smokers: a randomized controlled trial. Addiction. 2009 Nov;104(11):1891-900. doi: 10.1111/j.1360-0443.2009.02623.x. Epub 2009 Aug 28. PMID 19719796